CLINICAL TRIAL: NCT06227481
Title: Efficiency Of Combination Of Scar Subcision With Platelet Rich Plasma, Polydioxanone Mono Threads Or Fractional Carbon Dioxide Laser In The Treatment Of Severe Atrophic Acne Scars: A Randomized Controlled Study
Brief Title: Combined Procedures in the Treatment of Severe Acne Scars
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Omar Abdulrahman Hassan, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Severe acne scars
Record Dates: First submitted 2023-11-05; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Atrophic Acne Scar

STUDY DESIGN:
Intervention Model Description: This is a prospective controlled trial that will be conducted at Dermatology, venereology, and andrology Department, Al-Azhar university hospital, Assiut, in the period from December 2023 to December 2025, to assess the efficacy of combination of scar subcision with platelet rich plasma, polydioxanone mono threads or fractional carbon dioxide laserin the treatment of severe atrophic acne scars with 1:1:1 ratios and to compare between these modalities regarding safety and efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subcision plus platelet rich plasma (Active Comparator): 3 sessions of scar subcision with platelet rich plasma injection at the same session with one month interval
  Interventions: Procedure: Scar subcision; Procedure: Platelet rich plasma injection
- Subcision plus Polydioxanone mono threads (Active Comparator): 3 sessions of scar subcision followed by the insertion of Polydioxanone mono threads after the last session
  Interventions: Procedure: Scar subcision; Procedure: Polydioxanone mono threads insertion
- Subcision plus fractional carbon dioxide laser (Active Comparator): 3 sessions of scar subcision with Fractional carbon dioxide laser at the same session with one month interval
  Interventions: Procedure: Scar subcision; Device: Fractional carbon dioxide laser

INTERVENTIONS:
Procedure: Scar subcision — * Subcision will be performed with18 gauge cannula at the margin of the scars on both sides of the face.
  * The cannula will be directed in a forward and backward motion producing a tunnel. Then, the it will be passed in sideways in a sweeping action to freeing up the scars from their bases.
  * Once finish, the pressure will be applied to reduce the bleeding and swelling. The topical antibiotic will be applied for 3 days.
Procedure: Platelet rich plasma injection — • 20 ml of autologous whole blood will be collected into tubes containing acid citrate dextrose and centrifuged at 1500 rpm for 10 minutes in order to get PRP at the top of the test tube. Then, the PRP will be further centrifuged at 3700 rpm for 10 minutes at room temperature of 22°C in order to obtain a platelet count 4.5 times higher than the base line. Platelet-poor plasma (PPP) will be partly removed and partly used to resuspend the platelets. Calcium gluconate will be added as an activator (1:9), i.e., 1 ml of calcium gluconate in 9 ml of PRP
  Arms: Subcision plus platelet rich plasma
Procedure: Polydioxanone mono threads insertion — * Topical anesthetic cream will be applied for halfan hour on the involved area.
  * polydioxanone mono threads (50 mm, 27 G) will be inserted at 1-cm spacing into the dermal layer of the skin; the threads will be arranged in a transverse and vertical line in the form of a mesh similar to cross-hatching technique.
  * The total numbers will range from 8 to 10 each side. The skin of the face will be stretched by the non-dominant hand of the physician and the needle will be inserted by the other hand through the required point.
  Arms: Subcision plus Polydioxanone mono threads
Device: Fractional carbon dioxide laser — * Topical anesthetic cream will be applied for 30 minutes before the procedure.
  * BX300 device from AMI inc.,Korea will be used.
  * Different settings will be used according to each individual case regarding the type of scar, severity and skin type fluence ranging from 36 to 42 j/cm2 will be used and pulse duration 1.8 ms.
  * In an attempt to avoid common side effects that occur with fractional laser treatment, a lower fluence will be used in the first session and depending on the results, the fluence will be increased per treatment session.
  Arms: Subcision plus fractional carbon dioxide laser

SUMMARY:
Many methods utilize for acne scar treatment including laser, cosmetic filler, microneedling, local tumescent, Subcision and chemical peels. These procedures can be used individually or as a combination therapy.

Combining procedures give better results. In our study we will try in the period from March 2024 to March 2026, to assess the efficacy of combination of scar subcision with platelet rich plasma, Polydioxanone mono threads or fractional Carbon dioxide laser in the treatment of severe atrophic acne scars with 1:1:1 ratios and to compare between these modalities regarding safety and efficacy.

DETAILED DESCRIPTION:
This is a prospective controlled trial that will be conducted at Dermatology, venereology, and andrology Department, Al-Azhar university hospital, Assiut, in the period from March 2024 to March 2026, to assess the efficacy of combination of scar subcision with platelet rich plasma , polydioxanone mono threads or fractional carbon dioxide laser in the treatment of severe atrophic acne scars with 1:1:1 ratios and to compare between these modalities regarding safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

• Patients with severe atrophic acne scars (as per Goodman and Baron's acne qualitative scar grading scale)

Exclusion Criteria:

* Patients with active acne lesions.
* Patients having a keloid formation tendency.
* Patients with a history of bleeding disorder or severe anemia.
* Pregnant or lactating women.
* Patients received any treatment for scars in the last 6 months.
* Patients using drugs causing photosensitivity or systemic retinoids in the previous 6 months (for laser group).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Management of severe atrophic acne scars | 2 years
  to assess the efficacy of the combination of subcision with Platelet rich plasma, Polydioxanone mono threads or fractional carbon dioxide laser in the treatment of severe atrophic acne scars (As per Goodman and Baron's acne qualitative scar grading scale)

SECONDARY OUTCOMES:
Comparing the 3 lines | 2 years
  to compare between the combination of subcision with Platelet rich plasma, Polydioxanone mono threads or fractional carbon dioxide laser in the treatment of severe atrophic acne scars regarding efficacy and safety.
  (As per Goodman and Baron's acne qualitative scar grading scale)

CONTACTS AND LOCATIONS:
Overall Officials: Essam-Eldin M Mohamed, MD, Study Director — Al-Azhar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alser OH, Goutos I. The evidence behind the use of platelet-rich plasma (PRP) in scar management: a literature review. Scars Burn Heal. 2018 Nov 18;4:2059513118808773. doi: 10.1177/2059513118808773. eCollection 2018 Jan-Dec. PMID 30479843
- [Background] Chawla S. Split Face Comparative Study of Microneedling with PRP Versus Microneedling with Vitamin C in Treating Atrophic Post Acne Scars. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):209-12. doi: 10.4103/0974-2077.150742. PMID 25722599
- [Background] Chilicka K, Rogowska AM, Szygula R. Effects of Topical Hydrogen Purification on Skin Parameters and Acne Vulgaris in Adult Women. Healthcare (Basel). 2021 Feb 1;9(2):144. doi: 10.3390/healthcare9020144. PMID 33535651
- [Background] Goodman GJ, Baron JA. Postacne scarring: a qualitative global scarring grading system. Dermatol Surg. 2006 Dec;32(12):1458-66. doi: 10.1111/j.1524-4725.2006.32354.x. PMID 17199653
- [Background] Mu YZ, Jiang L, Yang H. The efficacy of fractional ablative carbon dioxide laser combined with other therapies in acne scars. Dermatol Ther. 2019 Nov;32(6):e13084. doi: 10.1111/dth.13084. Epub 2019 Oct 7. PMID 31496020
- [Background] Oh IY, Kim BJ, Kim MN. Depressed Facial Scars Successfully Treated with Autologous Platelet-Rich Plasma and Light-Emitting Diode Phototherapy at 830 nm. Ann Dermatol. 2014 Jun;26(3):417-8. doi: 10.5021/ad.2014.26.3.417. Epub 2014 Jun 12. No abstract available. PMID 24966653
- [Background] Zhang DD, Zhao WY, Fang QQ, Wang ZC, Wang XF, Zhang MX, Hu YY, Zheng B, Tan WQ. The efficacy of fractional CO2 laser in acne scar treatment: A meta-analysis. Dermatol Ther. 2021 Jan;34(1):e14539. doi: 10.1111/dth.14539. Epub 2020 Nov 23. PMID 33190373
- [Background] Nilforoushzadeh MA, Lotfi E, Heidari-Kharaji M, Nickhah N, Alavi S, Mahmoudbeyk M. Comparing cannula-based subcision with the common needle method: A clinical trial. Skin Res Technol. 2020 Jan;26(1):39-44. doi: 10.1111/srt.12761. Epub 2019 Aug 1. PMID 31373077
- [Background] Tan J, Beissert S, Cook-Bolden F, Chavda R, Harper J, Hebert A, Lain E, Layton A, Rocha M, Weiss J, Dreno B. Evaluation of psychological well-being and social impact of atrophic acne scarring: A multinational, mixed-methods study. JAAD Int. 2021 Dec 23;6:43-50. doi: 10.1016/j.jdin.2021.11.006. eCollection 2022 Mar. PMID 35005652